CLINICAL TRIAL: NCT02261844
Title: Resveratrol and Human Hepatocyte Function in Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No funding
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Brian G. Harbrecht, MD, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: ResveraCA
Record Dates: First submitted 2014-05-20; First posted 2014-10-10 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Liver Cancer
Keywords: Hepatocellular carcinoma; Metastatic colorectal cancer; Metabolism; Hepatic function
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular; Colorectal Neoplasms | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- resveratrol (Experimental): Resveratrol 1 g daily for 10 days
  Interventions: Dietary Supplement: Resveratrol
- Placebo (Placebo Comparator): Placebo 1 pill daily for 10 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Resveratrol — Resveratrol 1 gm po x 10 days prior to liver resection
  Other Names: Biotivia
  Arms: resveratrol
Drug: Placebo — Placebo 1 pill daily X 10 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if Resveratrol, a nutritional supplement, shows a beneficial effect in the cellular function of normal liver cells and diseased liver cells (cancer cells) in samples of liver tissue taken during elective liver surgery. Outcomes based on 3 measures will test the hypothesis that Resveratrol when used as a nutritional supplement will 1)improve metabolic function in liver cells, 2)reduce cellular growth and proliferation of cancer cells, 3)decrease inflammation in the liver.

DETAILED DESCRIPTION:
Hepatic function will be assessed by standard laboratory techniques. Hepatocyte signaling pathway proteins will be measured using western blot analysis for protein expression and polymerase chain reaction for gene expression. Activation of signaling pathways in both native hepatocytes and carcinoma will be analyzed by multi-plex signal array. The effect on transcription factors that may be important in gene expression will be analyzed by transcription factor array. The effect of resveratrol in altering hepatocyte and cancer cell metabolism will be analyzed by proteomic analysis.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective liver resection for liver cancer

Exclusion Criteria:

* Inability to speak or read English
* Sclerosing cholangitis, hemochromatosis, hepatic encephalopathy, acute hepatic failure
* History of daily alcohol intake
* Presence of human immunodeficiency virus
* Presence of significant renal dysfunction as defined by baseline serum creatinine > 2.0 mg/dl or need/impending need for chronic dialysis therapy
* Known allergy to the study medication
* Pregnancy, lactating women, women contemplating pregnancy during the study period

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Improved metabolic profile of liver cells | 36 months
  This outcome is a composite outcome and will be measured by assessing expression of multiple signaling proteins that are important in hepatic cell metabolism such as Akt, p38, Mitogen Activated Kinases, and Adenosine Monophosphate-activated Kinase (AMPK) and expression of gluconeogenic proteins such as Phosphoenolpyruvate carboxykinase (PEPCK).

SECONDARY OUTCOMES:
Decreased cell growth and proliferation | 36 months
  This outcome is a composite outcome of cellular pathways important in cancer cell replication. This will be measured by the expression of genes and proteins that regulate hepatic cell growth/cell survival such as cyclin gene expression, expression of the tumor suppressor p53, and expression of apoptosis proteins Bcl-2 and Bcl-xl.
Decreased hepatic inflammation | 36 months
  This outcome will be a composite outcome of pathways that regulate both cancer cell growth and inflammation. It will be measured by levels of genes and proteins for nitric oxide synthase, cytokines such as interleukin-6, and Nuclear Factor-kappa B signaling proteins.

CONTACTS AND LOCATIONS:
Overall Officials: Brian G Harbrecht, MD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States